CLINICAL TRIAL: NCT03056729
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single-Ascending-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BIIB076 in Healthy Volunteers and Subjects With Alzheimer's Disease
Brief Title: Single-Ascending-Dose Study of BIIB076 in Healthy Volunteers and Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 243HV101
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer's Disease; Healthy Volunteer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort HV1 (Experimental)
  Interventions: Drug: BIIB076; Drug: Placebo
- Cohort HV2 (Experimental)
  Interventions: Drug: BIIB076; Drug: Placebo
- Cohort HV3 (Experimental)
  Interventions: Drug: BIIB076; Drug: Placebo
- Cohort HV4 (Experimental)
  Interventions: Drug: BIIB076; Drug: Placebo
- Cohort HV5 (Experimental)
  Interventions: Drug: BIIB076; Drug: Placebo
- Cohort AD1 (Experimental)
  Interventions: Drug: BIIB076; Drug: Placebo

INTERVENTIONS:
Drug: BIIB076 — Administered as single intravenous (IV) infusion
Drug: Placebo — Administered as single IV infusion

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single-ascending intravenous (IV) infusions of BIIB076 in healthy volunteers and participants with Alzheimer's disease (AD). A secondary objective of the study for both healthy volunteers and participants with AD is to assess the serum pharmacokinetic(s) (PK) profile of BIIB076 after single-dose administration. Another secondary objective is to evaluate the immunogenicity of BIIB076 in serum after single-dose administration.

ELIGIBILITY:
Key Inclusion Criteria - Healthy Participants

* Must be in good health as determined by the Investigator, based on medical history and Screening evaluations.

Key Inclusion Criteria - Participants with Alzheimer's Disease (AD)

* Must meet all of the clinical criteria for mild cognitive impairment (MCI) due to AD or mild AD according to the National Institutes of Aging-Alzheimer's Association [McKhann 2011], and in addition must have the following:
* Clinical Dementia Rating (CDR) global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD.
* CDR Memory Box Score of ≥0.5.
* Mini-Mental State Examination score between 18 and 30 (inclusive) at Screening.
* Must have amyloid beta positivity confirmed at Screening

Key Exclusion Criteria - Healthy Participants

* Brain MRI findings that might pose a risk to the participant, or might prevent a satisfactory MRI assessment for safety monitoring.
* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Current enrollment in any other drug, biologic, device, or clinical study or treatment with an investigational drug or approved therapy for investigational use within 30 days (6 months for biologics) or 5 half-lives, whichever is longer, prior to Day-1.
* Contraindications to having a brain MRI (e.g., pacemaker; MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed).
* Contraindications to having an Lumbar Puncture (LP).

Key Exclusion Criteria - Participants with Alzheimer's Disease (AD)

* Any medical or neurologic/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause to the participant's cognitive impairment (e.g.,current history of substance abuse, uncontrolled vitamin B12 deficiency or uncontrolled thyroid disease, stroke or other cerebrovascular condition, Parkinson's disease, Lewy body dementia, or frontotemporal dementia or head trauma), or could lead to discontinuation, noncompliance with study assessments, or safety concerns.
* Diagnosis within 1 year prior to Screening and/or evidence of clinically significant (in the opinion of the Investigator) psychiatric illness including uncontrolled major depression, bipolar affective disorder, other psychiatric illness, and suicidal ideation.
* Any documented prior history of chronic schizophrenia.
* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary (including chronic obstructive pulmonary disease), neurologic, dermatologic, or renal disease, or other major disease, as determined by the Investigator.
* Use of any medications for the treatment of comorbid conditions that have not been stable for at least 8 weeks prior to Day -1 and/or that are not expected to remain stable for the duration of the study.
* Current enrollment or plan to enroll in any other drug, biologic, device, or clinical study or treatment with an investigational drug or approved therapy for investigational use within 30 days (6 months for biologics) or 5 half-lives, whichever is longer, prior to Day-1.
* Contraindications to having a brain MRI (e.g., pacemaker; MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed).
* Brain MRI findings that might be a contributing cause of the participant's dementia, might pose a risk to the participant, or might prevent a satisfactory MRI assessment for safety monitoring.
* Contraindications to having an LP.
* History of, or ongoing chronic uncontrolled hypertension
* History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class 3 or 4), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Day -1.
* Medications with platelet anti-aggregant or anticoagulant properties, except the use of aspirin at a dose ≤325 mg per day.
* For participants whose eligibility for study entry will be based on cerebral Aβ positivityas determined by amyloid PET (positron emission tomography), contraindication to having a PET scan (e.g., inability to lie flat or still for the duration of the scan) or intolerance to previous PET scans (i.e. previous hypersensitivity reactions to any PET radioligand or imaging agent, failure to participate in and comply with previous PET scans).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Week 20
  Safety surveillance

SECONDARY OUTCOMES:
BIIB076 serum pharmacokinetics (PK) concentration levels | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Area under the concentration-time curve from time zero to infinity (AUCinf) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Area under the concentration-time curve from time zero to the time of the last measurable sample (AUClast) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Maximum observed concentration (Cmax) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Time to reach maximum observed concentration (Tmax) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Terminal elimination half-life (t1/2) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Clearance (CL) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
PK parameter of BIIB076: Volume of distribution (Vd) | Up to Week 20
  Assessment of BIIB076 pharmacokinetics in blood
Number of participants with positive serum BIIB076 antibodies | Up to Week 20
  Serological assessment (of anti-BIIB076 antibodies in blood)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- United States (8):
  - MD Clinical, Hallandale, Florida
  - Bioclinica Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Indiana University, Indianapolis, Indiana
  - St Louis Clinical Trial, St Louis, Missouri
  - Covance Dallas CRU, Dallas, Texas
  - Covance CRU, Madison, Wisconsin